CLINICAL TRIAL: NCT02086097
Title: Effectiveness of Dexketoprofen Trometamol in the Management of Postoperative Endodontic Pain. Controlled Clinical Trial of Multiple Doses
Brief Title: Dexketoprofen Trometamol in Postoperative Endodontic Pain
Acronym: DTPEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Chavarría Bolaños (Other)
Responsible Party: Sponsor-Investigator, Daniel Chavarría Bolaños, Basic Sciences Laboratory, Dentistry School, Universidad Autonoma de San Luis Potosí
Organization: Universidad Autonoma de San Luis Potosí (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CEIFE-019-013
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Irreversible Pulpitis
Keywords: pain; symptomatic irreversible pulpitis; postoperative dental pain
MeSH Terms: conditions — Pain | interventions — dexketoprofen trometamol; Ibuprofen; 5'-palmitoyl cytarabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- dexketoprofen trometamol (Experimental): Administration of 25mg of Dexketoprofen Trometamol, 1 pill right after clinical procedure, the other 3 every 8 until the 24 hours administration period is completed
  Interventions: Drug: Dexketoprofen trometamol
- IBUPROFEN (Active Comparator): Administration of 600mg of Ibuprofen, 1 pill right after clinical procedure, the other 3 every 8 until the 24 hours administration period is completed
  Interventions: Drug: Ibuprofen
- PLACEBO (Placebo Comparator): 4 doses of sugar pills, 1 pill right after clinical procedure, the other 3 every 8 until the 24 hours administration period is completed
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Dexketoprofen trometamol — 25m of dexketoprofen (oral intake) every 8 hours
  Other Names: Miracox (Stein Labs); CODE: 00176101
  Arms: dexketoprofen trometamol
Drug: Ibuprofen — 600 mg of Ibuprofen (Oral Intake) every 8 hours
  Other Names: Ibuprofen Stein; CODE: 00065104
  Arms: IBUPROFEN
Drug: PLACEBO — INACTIVE SUGAR PILLS
  Other Names: PLAC
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to investigate the analgesic efficacy of multiple doses of Dexketoprofen Trometamol 25 mg on postoperative pain following emergency endodontic treatment in teeth with irreversible pulpitis, using as control Ibuprofen 600 mg and a placebo group.

Hypothesis:

Dexketoprofen trometamol when administered in multiple doses produces a greater effect to control postoperative pain after treating symptomatic irreversible pulpitis; in patients undergoing pulpotomy as an emergency procedure

DETAILED DESCRIPTION:
Pain management is an integral part of Endodontics, according to previously published results, pulp therapy and endodontic treatment induce postoperative pain more frequently than other dental procedures.

The prevalence of postoperative pain has been reported in 3-58% of cases, a positive association has been demonstrated between postoperative pain and the presence of apprehension and preoperative pain.

Although the incidence of moderate pain decreases within 1 day and substantially to minimal levels in 7 days after the endodontic treatment, severe postoperative pain occurs during the first 24 h.

Some drugs can prevent the production of inflammatory mediators involved in producing pain, such as prostaglandins.

Prostaglandin tissue levels are associated with patient reports of pain, and therefore, nonsteroidal anti-inflammatory drugs (NSAID's) may be key drugs for inflammatory pain abatement.

NSAIDs are widely available, and they have been reported to be effective in managing endodontic pain.

Ibuprofen is one of the most frequently used NSAIDs for control of postoperative pain associated with root canal treatment, and it has good efficacy and safety.

However an alternative treatment is Dexketoprofen Trometamol, a non-selective nonsteroidal anti-inflammatory drug, and a single isomer (S(+)-enantiomer) of ketoprofen formulated as trometamol salt. Dexketoprofen trometamol has been demonstrated to be effective in the treatment of acute pain.

The purpose of the study is assess the analgesic efficacy of multiple doses of Dexketoprofen Trometamol 25 mg on postoperative pain following emergency endodontic treatment in teeth with irreversible pulpitis This study was designed as a double-blind, randomised, placebo-controlled clinical trial. Following the guidelines suggested by CONSORT group for planning and reporting clinical trials. The ethics committee of the faculty of Dentistry approved the study design. All of the subjects will be informed of the possible risk of endodontic therapy and experimental treatments and will sign institutionally approved consents forms.

In total, 87 patients will be included in this study. The simple size calculation was performed with a type error of 0.05 and statistical power of 80% on the basis of report of the analgesic efficacy of Dexketoprofen Trometamol 25 mg vs Ibuprofen 600 mg after their administration in patients subject to oral surgery.

All of the subjects voluntarily will presented at the postgraduate endodontics clinic of the Faculty of Dentistry at San Luis Potosí University. The select subjects will have a diagnosis of symptomatic irreversible pulpitis.

Pain will be scored using numerical rating scale, this is a 11 point scale where the end points are the extremes of no pain and pain as bad as it could be, or worst pain. Accordingly, no pain corresponded with 0, mild pain with 1-3, moderate pain with 4-6, and severe pain 7 and above.7 After the endodontic emergency treatment, patients will be randomly divided into three groups of 27 patients each. A control group will receive multiple doses of placebo and 2 experimental groups receive multiple dose of ibuprofen (600 mg) and Dexketoprofen trometamol (25 mg). The first dose of medication is given once the procedure is completed, the following doses will be taken every 8 hours to cover a total of 24 hours.

Patients will be monitored to assess the therapeutic effect at different time intervals, 1,8,16,24,48 and 72 hours using numerical rating scale.

If the analgesic efficacy is not achieved Supradol (Ketorolac 30 mg) or Zaldiar (Paracetamol 325mg/Tramadol 37.5 mg) will be taken as rescue medication.Any adverse events or symptoms will be recorded.

Statistics Normal distribution will be tested by the Student's-t test or mann-whitney U test. A non -parametric chi-squared test was performed to identify statistically significant differences between the groups; the level of significance was set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years and older with moderate-to-severe dental pain assessed by numerical rating scale (NRS) associated with irreversible pulpitis.

Exclusion Criteria:

* • Female pregnant or breastfeeding

  * Used pain relievers or anti-inflammatory drugs within 24 hours preceding emergency endodontic treatment
  * Have any significant medical condition
  * Taking any medications for anxiety, depression or schizophrenia
  * Have a history of hypersensitivity to nonsteroidal anti-inflammatory drugs (NSAIDs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
post operative pain measurement in symptomatic irreversible pulpitis, after multiple doses of dexketoprofen trometamol | 1 observation after 72 hours of emergency clinical procedure (Pulpotomy) for pain management
  Using a visual analogue scale, each patient is asked to inform the researcher team about postoperative pain levels at 1, 8, 16, 24, 48 and 72 hours after pulpotomy procedure as emergency clinical manage of endodontic pain in irreversible pulpitis cases. Patients will be asked to take multiple doses of either Dexketoprofen Trometamol 25mg, Ibuprofen 600mg or placebo pills. Also, aspects like local anesthetic effect duration and local/systemic side effects will be monitored. Each patient will have a personal file to record the information during each period (1, 8, 16, 24, 48 and 72 hours )

SECONDARY OUTCOMES:
Duration of the activity of the analgesic treatment | observation periods of 1, 8, 16, 24, 48 AND 72 hours
  The duration of the effect of each drug will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Rodríguez, DDS, Principal Investigator — Universidad Autonoma San Luis Potosi; Amaury J Pozos-Guillen, PhD, Study Chair — Universidad Autonoma San Luis Potosi; Daniel Chavarria, PhD, Study Director — Universidad Autonoma San Luis Potosi
Locations (1):
- Endodontics Master Degree program, Dentistry Faculty, San Luis Potosi University, San Luis Potosí City, San Luis Potosí, Mexico